CLINICAL TRIAL: NCT05489757
Title: SPY Portable Handheld Imaging (SPY-PHI) System With SPY-QP Software for Quantitative Fluorescence Angiography With IndoCyanine Green for Perfusion Assessment During Surgery
Brief Title: Quantitative Fluorescence Angiography With ICG for Perfusion Assessment During Surgery
Acronym: SPY Q-ICG PAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Lorenzo Cinelli, Clinical Research Fellow, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 154/INT/2021
Record Dates: First submitted 2022-06-24; First posted 2022-08-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Esophagus; Fistula; Fistula;Rectal; Complication of Surgical Procedure; Complication,Postoperative
Keywords: ICG quantification; Esophagectomy; Colorectal resection; Perfusion assessment
MeSH Terms: conditions — Esophageal Fistula; Rectal Fistula; Postoperative Complications | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Prospective, Interventional, Monocentric Cohort Study on Medical Device (CE marked, according to indications for use) Prospective, Observational, Monocentric, Pharmacologic Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SPY Portable Handheld Imaging (SPY-PHI) System with SPY-QP Software — Perfusion assessment with SPY Q-ICG system

SUMMARY:
The accurate assessment of intraoperative tissue perfusion is essential in any branch of surgery. Anastomotic leakage (AL) is one of the most feared complications following gastrointestinal surgery, with potentially threatening consequences resulting in worsened short- and long-term outcomes. Consistently, a recent meta-analysis showed a correlation between AL and shorter disease-free survival in colorectal surgery. Despite its multifactorial origin, AL is highly related to inadequate visceral perfusion. Traditionally, perfusion assessment and subsequent anastomotic viability have been evaluated by surgeons using intraoperative indicators, such as color, pulsation of vessels, presence of peristalsis and bleeding from the resection lines. However, these clinical parameters are not able to reliably assess the real visceral perfusion and their evaluation is limited in minimally invasive surgery. Hence, the growing interest for innovative techniques able to properly assess tissue perfusion. Among these, the fluorescence angiography (FA) with indocyanine green (ICG) has become increasingly popular during the last decade, although its approval for biomedical purposes by the Food and Drug Administration (FDA) dates back to 1956. ICG is an amphiphilic, non-toxic, tricarbocyanine iodide dye that can be safely injected intravenously and is exclusively eliminated by the liver, without any absorption. Thanks to its fluorescent properties, it allows the real-time visualization of tissue vascularization. FA with ICG has shown promising results for the evaluation of perfusion in numerous surgical procedures, thus leading to modifications of the surgical strategy and consequently to a decrease in the rates of AL. On the other hand, ICG interpretation is subjective, based on the evaluation of fluorescence performed by the operating surgeon. These results lack into a high inter-observer variability and affect the possibility to obtain objective, reproducible and reliable tissue perfusion assessments.

Quantitative fluorescence angiography with ICG (Q-ICG) could overcome these limitations. In Q-ICG the fluorescence signal is elaborated by a new computer quantification algorithm and translated into a fluorescence-time curve (FTC), from which several Q-ICG parameters and values can be extracted. Given the power of ICG in reflecting the perfusion of examined tissues, a new quantification algorithm has the potential to turn the subjective parameters derived from surgeon's perspective into objective numeric values.

The primary aim of this study is to evaluate which Q-ICG values provided by a new quantification algorithm correspond to subjective perfusion parameters usually evaluated by the surgeon in patients undergoing left colon, rectal or esophagogastric resections.

The secondary aim is to evaluate possible correlations between Q-ICG values provided by the quantification algorithm and perioperative outcomes.

DETAILED DESCRIPTION:
The study is designed as a prospective, observational, monocentric, cohort study on algorithm. At our Institution ICG is already used routinely to assess visceral perfusion during gastrointestinal operations. We plan to enroll 70 patients for esophagogastric resections and 140 patients for colorectal resections. Firstly, the adequacy of colon or gastric perfusion will be assessed by the surgical team in the traditional way. Color, pulsatile flow of vessels (right gastroepiploic arcade for the gastric conduit, marginal artery for the colon), presence of peristalsis and bleeding from the colic resection lines will be considered as parameters of perfusion. Then, ICG will be injected, Q-ICG analysis will be performed in all the patients by using a new quantification algorithm and data will be recorded and reported in a specific Database. The surgical strategy will not be modified based on Q-ICG results.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to give informed consent for participation in the trial
* Male and Female, Age > 18 years
* Patients undergoing left colon, rectal or esophagogastric resections
* Patients with malignant or benign disease
* Minimally invasive or open approach surgery

Exclusion Criteria:

* Absence of esophagogastric or colorectal reconstruction (e.g. Miles procedure)
* Limited sigmoid resection without ligation of the inferior mesenteric artery
* Known allergies, hypersensitivity or intolerance to indocyanine green (ICG) or iodine contrast agents,
* Patients with hyperthyroidism or benign thyroid tumor
* Acute or chronic kidney failure (stage ≥ 3)
* Pregnant or lactating women, or with a positive pregnancy test performed before surgery
* Any clinical condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum intensity of ICG fluorescence | One timepoint: at day 0, after the externalization of colon/stomach, before packing the colorectal/esophagogastric anastomosis.
  % (absolute value)
Time to first ICG fluorescence signal | One timepoint: at day 0, after the externalization of colon/stomach, before packing the colorectal/esophagogastric anastomosis.
  seconds
Time-to-peak | One timepoint: at day 0, after the externalization of colon/stomach, before packing the colorectal/esophagogastric anastomosis.
  seconds

SECONDARY OUTCOMES:
Correlation with postoperative outcomes | From day 0 to day 30 after discharge
  The rate of anastomotic leakage in patients who underwent colorectal or esophagogastric resections

CONTACTS AND LOCATIONS:
Locations (1):
- Lorenzo Cinelli, Milan, Italy

IPD SHARING:
Plan to Share IPD: No